CLINICAL TRIAL: NCT03766893
Title: Comparing Medication Maintenance in Comprehensive Community and Pharmacy Settings to Enhance Engagement
Brief Title: Medication Maintenance Therapy in Community Pharmacy Settings
Acronym: MATPharm
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Traci Green, Senior Research Scientist, Associate Professor of Emergency Medicine, Lifespan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1112133
Record Dates: First submitted 2018-10-02; First posted 2018-12-06 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacy based opioid use disorder care (Experimental): A single-arm pilot study to test the collaborative pharmacy practice agreement for MAT (using the medications buprenorphine or injectable naltrexone) care model with up to 12 patients with opioid use disorder, assessing feasibility of medication dispensing, administration, and monitoring in the pharmacy, and determining patient acceptability of this model.
  Interventions: Drug: Buprenorphine / Naloxone Oral Product; Drug: injectable naltrexone; Other: Pharmacy maintenance addiction care

INTERVENTIONS:
Drug: Buprenorphine / Naloxone Oral Product — To treat opioid use disorder, buprenorphine/naloxone will be provided by a study pharmacist under a collaborative pharmacy practice agreement on a weekly (buprenorphine/naloxone) basis, unless the care plan specifies greater frequency of pharmacy visit. The median expected dose of buprenorphine/naloxone (sublingual film or tablet) is 8 to 24 mg daily, and may be adjusted per the collaborative pharmacy practice agreement.
Drug: injectable naltrexone — To treat opioid use disorder, injectable naltrexone will be provided by a study pharmacist under a collaborative pharmacy practice agreement on a monthly (injectable naltrexone) basis. The expected dose of injectable naltrexone will be approximately 380 mg. Injectable naltrexone will be dispensed and prepared by the pharmacist but administered by nursing staff for the pilot study.
Other: Pharmacy maintenance addiction care — Patients on a stable dose of buprenorphine/naloxone or naltrexone will receive maintenance care at the pharmacy for one month. Patients will visit weekly for check-ins with a pharmacist. Patients on buprenorphine/naloxone will be dispensed their medication at study visits, whereas patients taking injectable naltrexone will be dispensed it once by the pharmacist during the pilot. All patients will visit the pharmacy at least weekly for addiction care (assessment, toxicological testing).

SUMMARY:
The goal of this study is to examine how the pharmacy can better optimize treatment expansion by providing pharmacy-based medication assisted treatment (MAT) for maintenance under a collaborative pharmacy practice agreement.

DETAILED DESCRIPTION:
This study will be the first to develop and use a collaborative pharmacy practice agreement (CPA) for medication assisted treatment (MAT) intended for statewide application. This will also be the first study to use a randomized controlled trial design to test the multisite implementation of known effective interventions to treat opioid use disorder and prevent fatal opioid overdose (treatment with buprenorphine and natlrexone) in a pharmacy setting. Understanding how this model can improve engagement in care within innovative systems of MAT delivery like the Rhode Island Centers of Excellence in MAT model as well as the more traditional office based opioid therapy (OBOT) arrangement, and for patients with shorter and longer time on stabilized MAT doses advances the science of addiction health services.

This study presents an opportunity to compare clinical outcomes of patients randomized to receive the same medications but in different settings that are equipped with differing levels of counseling expectations and access to wrap-around services. In this way, the trial helps to inform whether-and for whom--the limited support services in the pharmacy are sufficient to engage and retain patients in MAT, or if ready access to comprehensive services are necessary. Approximately 86% of Americans live within 5 miles of a pharmacy, making pharmacists the most accessible health care professionals. This model could redefine the role of the pharmacy.

The initial phase of the study (Phase 1) involves preparation for and conduct of a pilot study of the pharmacy MAT care model.

The aims of the first study phase (R21 grant) are:

* Aim 1: Develop a pharmacy CPA for the management of opioid use disorder using buprenorphine and naltrexone.
* Aim 2: For patient inmates maintained at the Rhode Island Department of Corrections, assess the feasibility and timing of randomization and transfer to a CPA pharmacy providing MAT post-release. This targeted assessment will inform the R33 design.
* Aim 3: Pilot test the pharmacy MAT model with up to 12 patients, assessing feasibility of medication dispensing, administration, and monitoring in the pharmacy, and determining patient acceptability of this model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* English speaking; currently enrolled at a CODAC site in Rhode Island for the treatment of opioid use disorder;
* maintained on a stable dose of buprenorphine or injectable naltrexone for at least 2 days;
* no stable co-morbid illnesses likely to progress clinically during the pilot study;
* able and willing to provide written informed consent and locator information (working telephone and >2 contacts) to participate.

Exclusion Criteria:

* currently pregnant or trying to get pregnant;
* plans to move or leave the state during the study, including pending legal action;
* self reported past year suicide attempt or self-reported past year suicidal thoughts with a plan;
* any condition that, in the researchers' judgment, interferes with safe study participation or adherence to study procedures, including but not limited to a mental, medical or other substance use disorder that is likely to require ongoing, intense clinical management during the pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacists' dispensing of MAT medications | up to one month
  Measured by the number of MAT medications dispensed from a study pharmacy according to the pharmacy records, over the one month pilot period.
Pharmacists' monitoring of MAT care | up to one month
  Measured by the number of toxicological drug screens performed at a study pharmacy over the one month pilot period.
Pharmacist-reported feasibility of executing the collaborative pharmacy practice: agreement for MAT: Likert scale | up to one month
  7-point Likert scale item assessing the pharmacist's view of the overall model feasibility. The item asks: How acceptable is providing buprenorphine/Suboxone care at the pharmacy?
  With responses ranging from 1 to 7 as:
  1. totally unacceptable
  2. unacceptable
  3. slightly unacceptable
  4. neutral
  5. slightly acceptable
  6. acceptable
  7. perfectly acceptable
  Higher scores represent better outcome (i.e., endorsement of acceptability of the model), according to the pharmacists.
Patient acceptability of pharmacy-provided MAT care: Likert scale | up to one month
  7-point Likert scale item assessing overall acceptability of the pharmacy MAT model. The item asks: How acceptable is going to the pharmacy for your buprenorphine/Suboxone care? With responses ranging from 1 to 7 as:
  1. totally unacceptable
  2. unacceptable
  3. slightly unacceptable
  4. neutral
  5. slightly acceptable
  6. acceptable
  7. perfectly acceptable
  Higher scores represent better outcome (i.e., high endorsement of acceptability of the model), according to the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Traci C Green, Principal Investigator — Lifespan
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States